CLINICAL TRIAL: NCT01717105
Title: Observational Post-authorization Prospective Study to Characterize the Incidence of Epidermal Growth Factor Receptor (EGFR) Mutation Positive and Advanced Non-small Cell Lung Cancer Patients and Their Clinical Management in Galicia
Brief Title: Observational Study to Characterize the Incidence of EGFR Mutation Positive and Advanced NSCLC Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Grupo Gallego de Cancer de Pulmon (Other)
Collaborators: AstraZeneca (Industry); Dynamic Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: GGCP 048-10; GGC-CPN-2010-01 (Other: AEMPS)
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Metastatic Non-Small-Cell Lung Cancer
Keywords: Non-small cell lung cancer (NSCLC); Epidermal growth factor receptor (EGFR) positive mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Tumor tissue Plasma samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- metastatic non-small cell lung cancer: Only epidermal growth factor receptor (EGFR) M+ patients will be eligible for the study assessments

SUMMARY:
The present study has been designed in order to characterize the incidence of patients with advanced non-small cell lung cancer (NSCLC) carrying epidermal growth factor receptor (EGFR) positive mutations and their clinical management in Galicia.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for patients´ screening:

* Patients of both sexes aged 18 or more.
* Histologically confirmed advanced or metastatic Non-Small-Cell Lung Cancer (NSCLC) (patients stage III B unsuitable for locoregional treatment, and stage IV).
* Chemo- naïve patients (Non-Small-Cell Lung Cancer patients who have not received first line systemic cytotoxic chemotherapy).
* Patients with available tumoral tissue (primary tumor or metastatic area) or cytological samples including fine needle aspirates (primary tumor or metastatic area), bronchial alveolar lavage or bronchial scrapings and pleural effusion.
* Patients who have granted their written informed consent.

Patients must fulfill the inclusion criteria previously mentioned and the following one in order to be enrolled in the study (visit 1) for the follow-up until progression or until 9 months from the beginning of treatment have elapsed:

Inclusion Criteria for patients´ follow-up

* Patients with documented positive mutation in epidermal growth factor receptor (EGFR) (M+).

Exclusion Criteria:

* Combined histology of non-small cell and small cell lung cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient consultation in oncology
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-12 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients with epidermal growth factor receptor (EGFR) positive mutation among advanced or metastatic non-small-cell lung cancer (NSCLC) patients in Galicia | 10 months (recruitment period)

SECONDARY OUTCOMES:
Epidermal growth factor receptor (EGFR) mutational status in tumor tissue (primary tumor or metastatic samples) and plasma samples at screening | 1 day (Screening Visit)
Type of epidermal growth factor receptor (EGFR) mutations: deletion in exon 19, point mutation at codon 858 (L858R) or other (only for EGFR M+ patients) | 1 day (Screening Visit)
Prescribed first line treatment (only for epidermal growth factor receptor (EGFR) M+ patients) | 1 day (First study visit)
Tumor response (only for epidermal growth factor receptor (EGFR) M+ patients) | From inclusion until disease progression, death or until 9 months from the inclusion of the last patient in the study have elapsed, whichever is earlier.
Disease control (only for epidermal growth factor receptor (EGFR) M+ patients) | From inclusion until the end of the study (9 months subsequent to the last patient's inclusion or until lost of follow-up)
Prescribed second-line treatment after progression (only for epidermal growth factor receptor (EGFR) M+ patients) | 1 day (Progression Visit)
Progression-free survival and overall survival (only for epidermal growth factor receptor (EGFR) M+ patients) | 1 day (at the end of the study 9 months subsequent to the last patient's inclusion or until lost of follow-up
Epidermal growth factor receptor (EGFR) mutational status at disease progression in tumor tissue (primary tumor or metastatic samples) and plasma samples (only for EGFR M+ patients) | 1 day (Progresion Visit)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Vázquez Estévez, Doctor, Study Director — Grupo Gallego de Cáncer de Pulmón (GGCP)
Locations (9):
- Spain (9):
  - Centro Oncologico de Galicia, A Coruña, A Coruña
  - Complexo Hospitalario Arquitecto Marcide, Ferrol, A Coruña
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Lucus Augusti Hospital, Lugo, Lugo
  - Complejo Hospitalario de Ourense, Ourense, Orense
  - Complexo Hospitalario de Pontevedra, Pontevedra, Pontevedra
  - Hospital do Meixoeiro, Vigo, Pontevedra
  - Hospital Xeral-Cíes, Vigo, Pontevedra
  - Hospital Povisa, Vigo, Pontevedra